CLINICAL TRIAL: NCT05746078
Title: Long-term Assessment of the Performance and Safety of SPRING THREAD® Elastic Tensor Thread.
Brief Title: Performance and Safety Assessment of SPRING THREAD® Elastic Tensor Thread in Patients with Mild to Moderate Facial Ptosis.
Acronym: ESTES
Status: Recruiting | Type: Observational
Sponsor: 1st SurgiConcept (Industry)
Collaborators: EVAMED (Other)
Responsible Party: Sponsor
Other Study IDs: ESTES
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Ptosis; Ptosis, Mild
Keywords: Ptosis, Moderate
MeSH Terms: conditions — Blepharoptosis; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this post-market clinical follow up study is to assess the safety and effectiveness of the SPRING THREAD® elastic tensor thread. The study will evaluate the outcome of the SPRING THREAD® elastic tensor thread range over a period of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Men / women aged 35 to 75 with facial ptosis (cheekbones, jowls) with or without a history of aesthetic treatment (botox, filler, surgical lift).
* Patient able to understand the explanations given.
* Patient informed and not objecting to participate in the study.
* Patient able to comply with protocol requirements, including follow-up visits.
* Patient affiliated to social security.

Exclusion Criteria:

* Patient unable to understand study information and attend study visits.
* Patient did not give consent to participate.
* Patients who have had a previous facial rejuvenation treatment in the 3 months prior to the study.
* Patients treated with long-term systemic corticosteroids.
* Patients with visceral failure, chronic immunological pathology, pregnant or breasfeading women.
* Patient participating or having participated in another clinical trial protocol, drug or medical device within 30 days of inclusion.
* Patient refusing to participate in the clinical investigation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population involved are men or women aged 35 to 75 with facial ptosis (mild to moderate) eligibles for tensor thread treatment.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2023-02-16 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Investigator Global Aesthetic Improvement Scale (IGAIS) | At 12 months
  Proportion of patients with an IGAIS score between 1 and 3 showing an improvement of ptosis.
  This item is scaled from 1 to 5, 5 being the worst value.

SECONDARY OUTCOMES:
Patient satisfaction with SGAIS score (Subject Global Aesthetic Improvement Scale) | Day 0 to Year 5.
  The patient satisfaction with SGAIS score will be assessed at each visit. This item is scaled from 1 to 5, 5 being the worst value.
Surgeon satisfaction with IGAIS score (Investigator Global Aesthetic Improvement Scale) | Day 0 to month 24
  The surgeon satisfaction with the IGAIS score will be assessed from intervention (day 0) to 12 months.
  This item is scaled from 1 to 5, 5 being the worst value.
Improvement of overall facial appearance | Day 0 to Year 5.
  The improvement of overall facial appearance (harmony) will be assessed using a 5-point patient satisfaction scale.
  The worst value is very unsatisfied and the highest value is very satisfied.
Age of face | Day 0 to year 5.
  The age of patient face will be assessed a specific question at each visit.
Safety of SPRING THREAD® Elastic Tensor Thread | Day 0 to month 12.
  All adverse event will be assessed for the study duration.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Henri Mondor, Créteil
  - Hôpital Pierre Paul Riquet, Toulouse